CLINICAL TRIAL: NCT03361982
Title: Randomized Controlled Trial Comparing Fresh Vs Frozen Surgical Sperm in In Vitro Fertilization Cycles
Brief Title: Fresh Vs Frozen Surgical Sperm in IVF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment issues
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RMA-2017-06
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresh surgical testicular sperm (No Intervention): Fresh, surgically obtained testicular sperm
- Frozen surgical testicular sperm (Experimental): Surgically obtained testicular sperm that will undergo slow freezing and thawing
  Interventions: Other: Slow Freezing and Thawing

INTERVENTIONS:
Other: Slow Freezing and Thawing — half of the surgically obtained testicular sperm will be frozen for 30 minutes and subsequently thawed prior to performing ICSI
  Arms: Frozen surgical testicular sperm

SUMMARY:
The primary objective of this study is to determine if the use of frozen surgical testicular sperm specimens for ICSI lead to different IVF outcomes when compared with the use of fresh surgical testicular sperm for ICSI.

DETAILED DESCRIPTION:
The study seeks to isolate the effect of slow freezing and thawing of surgical sperm specimens on fertilization and embryo blastulation rates by utilizing a randomized controlled split cohort protocol including men with obstructive azoospermia undergoing surgical sperm retrieval and good-prognosis female patients.

ELIGIBILITY:
Inclusion Criteria:

* Females age < 42 with an indication for IVF
* Females with lowest AMH level 1.2 ng/mL or higher
* Females with FSH < 13 mIU/mL
* Sperm obtained via Surgical retrieval (any type) for IVF only
* Use of comprehensive chromosome screening (CCS) to screen embryos for aneuploidy
* BMI < 35
* Baseline antral follicle count of > 8
* Single embryo transfers only

Exclusion Criteria:

* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.
* Contraindication to IVF
* Clinical indication for preimplantation genetic diagnosis (PGD) (i.e., screening for single gene disorder, chromosomal translocation, or any other disorders requiring detailed embryo genetic analysis)
* Fewer than 4 mature oocytes retrieved (will not randomize)
* Male partner with non-obstructive azoospermia
* Male partner with any Karyotype other than 46,XY
* Male partner with history of spinal cord injury
* Male partner with Kallman's syndrome
* History of chronic oligomenorrhea
* History of hydrosalpinges or adnexal mass
* History of endometrial insufficiency (max endometrial thickness < 7mm)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Blastulation Rate | 5-7 days post ICSI procedure
  total number of embryos reaching the blastulation stage of development

SECONDARY OUTCOMES:
Fertilization Rate | 1 day post ICSI
  number of 2PNs
Time to Find Sperm in Fresh Specimen | up to 6 hours post surgery
  total amount of time spent finding sperm in the fresh surgical testicular sperm sample
Post-thaw recovery rate of frozen surgical sperm | 30 minutes after freezing
  analysis of sperm parameters post freezing
Aneuploidy Rate | 2 weeks post trophectoderm biopsy
  number of chromosomally normal and abnormal embryos
Implantation Rate | approximately 4-6 weeks post embryo transfer
  presence of fetal heart beat at discharge to obstetric care

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Tiegs, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine LA, Dimitriou RJ, Fakouri B. Testicular and epididymal percutaneous sperm aspiration in men with either obstructive or nonobstructive azoospermia. Urology. 2003 Aug;62(2):328-32. doi: 10.1016/s0090-4295(03)00374-1. PMID 12893345
- [Background] Cui X, Ding P, Gao G, Zhang Y. Comparison of the Clinical Outcomes of Intracytoplasmic Sperm Injection Between Spermatozoa Retrieved From Testicular Biopsy and From Ejaculate in Cryptozoospermia Patients. Urology. 2017 Apr;102:106-110. doi: 10.1016/j.urology.2016.08.071. Epub 2016 Nov 25. PMID 27894976
- [Background] Ben-Ami I, Raziel A, Strassburger D, Komarovsky D, Ron-El R, Friedler S. Intracytoplasmic sperm injection outcome of ejaculated versus extracted testicular spermatozoa in cryptozoospermic men. Fertil Steril. 2013 Jun;99(7):1867-71. doi: 10.1016/j.fertnstert.2013.02.025. Epub 2013 Mar 13. PMID 23490166
- [Background] Pabuccu EG, Caglar GS, Tangal S, Haliloglu AH, Pabuccu R. Testicular versus ejaculated spermatozoa in ICSI cycles of normozoospermic men with high sperm DNA fragmentation and previous ART failures. Andrologia. 2017 Mar;49(2). doi: 10.1111/and.12609. Epub 2016 Apr 25. PMID 27108915
- [Background] Ohlander S, Hotaling J, Kirshenbaum E, Niederberger C, Eisenberg ML. Impact of fresh versus cryopreserved testicular sperm upon intracytoplasmic sperm injection pregnancy outcomes in men with azoospermia due to spermatogenic dysfunction: a meta-analysis. Fertil Steril. 2014 Feb;101(2):344-9. doi: 10.1016/j.fertnstert.2013.10.012. Epub 2013 Dec 9. PMID 24345355
- [Background] Forman EJ, Li X, Ferry KM, Scott K, Treff NR, Scott RT Jr. Oocyte vitrification does not increase the risk of embryonic aneuploidy or diminish the implantation potential of blastocysts created after intracytoplasmic sperm injection: a novel, paired randomized controlled trial using DNA fingerprinting. Fertil Steril. 2012 Sep;98(3):644-9. doi: 10.1016/j.fertnstert.2012.04.028. Epub 2012 May 17. PMID 22608316